CLINICAL TRIAL: NCT06577545
Title: Design, Implementation and Evaluation of a Behavioural Intervention to Treat Obesity in Breast Cancer Survivors.
Brief Title: Lifestyle Behavioural Intervention on Breast Cancer Survivors for the Treatment of Overweight/Obesity.
Acronym: Nutri-Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Odysseas Androutsos, Professor of Nutrition and Clinical Dietetics, Department of Nutrition and Dietetics, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Behavioral Intervention in BCS
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer Female; Overweight and Obesity
Keywords: behavioural intervention; lifestyle intervention; nutrition and physical activity; breast cancer survivors; overweight and obesity; digital counselling
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (UC) (No Intervention): Participants in Usual Care (UC) study arm will receive WCRF cancer prevention recommendations.
- Behavioural Lifestyle (BL) (Active Comparator): 24-week behavioural lifestyle intervention program.
  Interventions: Behavioral: Behavioural Lifestyle (BL)

INTERVENTIONS:
Behavioral: Behavioural Lifestyle (BL) — 24-week behavioural lifestyle intervention
  Arms: Behavioural Lifestyle (BL)

SUMMARY:
The goal of this clinical trial is to compare a behavioural lifestyle intervention program (BL) to usual care (UC) in breast cancer survivors. The main questions it aims to answer are:

1. If the participants of the BL group will lose more weight than the UC group.
2. If the participants of the BL group will have more lifestyle benefits than the UC group.

Volunteers will participate in a 24-week behavioural program. This program aims to improve their nutrition and physical activity in order to lose at least 10% of their initial body weight.

DETAILED DESCRIPTION:
Eligible participants should be female breast cancer survivors between the ages of 18 and 65, with a BMI between 25 and 40 kg/m2, and no active cancer therapy or ongoing treatment, except for hormonal or immune therapy.

The usual care (UC) group will receive WCRF cancer prevention recommendations. The behavioural lifestyle intervention program (BL) group will participate in a 24-week intervention targeting diet and physical activity to lose weight.

The program will be considered successful if participants lose at least 10% of their initial body weight. A secondary goal is to improve their nutrition and physical activity levels. The third and last goal is to improve their overall quality of life and their anxiety levels.

The behavioral program includes in-person online meetings, group online sessions, and digital counseling material. Considering that participants will be residing all around Greece, an internet videoconferencing technology will be required.

A qualitative study incorporating focus groups undertaken prior to this study to establish the methodology resulted in the utilization of synchronous and asynchronous media, as well as a combination of in-person and group sessions.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 40 kg/m2

Exclusion Criteria:

* active cancer or any ongoing treatment except hormonal or immune therapy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study includes only biological female participants
Enrollment: 92 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
body weight change | From enrollment to the end of treatment at 24 weeks
  % of the initial body weight change

CONTACTS AND LOCATIONS:
Overall Officials: Odysseas Androutsos, Professor, Study Chair — University of Thessaly
Locations (1):
- University of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: Researchers under request

REFERENCES:
- [Background] Perperidi M, Saliari D, Christakis C, Huybrechts I, Saloustros E, Theodorakis Y, Androutsos O. Identifying the effective behaviour change techniques in nutrition and physical activity interventions for the treatment of overweight/obesity in post-treatment breast cancer survivors: a systematic review. Cancer Causes Control. 2023 Aug;34(8):683-703. doi: 10.1007/s10552-023-01707-w. Epub 2023 May 6. PMID 37149509
- [Background] Perperidi M, Saltaouras G, Konstandis A, De Craemer M, Saloustros E, Theodorakis Y, Androutsos O. Barriers and facilitators of healthy lifestyle and perspectives towards the development of weight loss programmes. Focus groups with post-treatment breast cancer survivors in Greece. J Nutr Sci. 2023 Nov 3;12:e111. doi: 10.1017/jns.2023.94. eCollection 2023. PMID 37964978
- [Background] Saltaouras G, Perperidi M, Vantzou D, Vatsina K, Saloustros E, Theodorakis Y, Androutsos O. Determinants of lifestyle and body weight status among breast cancer survivors with overweight/obesity and perspectives towards the development of weight loss interventions: a qualitative study with health professionals from Greece. J Nutr Sci. 2024 Jan 23;13:e4. doi: 10.1017/jns.2023.117. eCollection 2024. PMID 38282654